CLINICAL TRIAL: NCT07118826
Title: Evaluation and Refinement of a Trauma-Informed and Peer Supported Mobile Brief Intervention for Young Adult Substance Users With Interpersonal Trauma
Brief Title: A Brief Intervention for Young Adult Substance Users With Interpersonal Trauma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western Kentucky University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1839376-8
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Heavy Drinking; Alcohol Drinking; Substance Use; Drinking Behavior
Keywords: Brief intervention; Alcohol; Trauma; Drinking; Peer coaching
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders; Drinking Behavior; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either 1) a standard brief intervention 2) a modified brief intervention with peer coaching and trauma-related information
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Brief Intervention (Experimental): Immediately following completion of the baseline assessment, participants will be texted a link to a secure website which contains the participant's personalized feedback. Personalized feedback is automatically presented via a programming algorithm that is based on the participants baseline survey responses. The personalized feedback component will include a personalized substance use profile, information on peer norms, prior substance-related consequences experienced by the participant, practical costs (e.g., money spent on substances, fees for a DUI), and standard protective behavioral strategies to limit substance-related risk.
  Interventions: Behavioral: Standard Brief Intervention; Behavioral: Trauma-Informed and Peer-Supported Brief Intervention
- Trauma-Informed and Peer-Supported Brief Intervention (Experimental): In addition to the components of the standard brief intervention, the TIPS-BI will include personalized feedback about participants use of substances to cope. Additionally, participants will be provided with psychoeducation about the link between substance use, trauma, and coping motives, and information highlighting the iatrogenic effects that substance use has on negative emotions. Participants will also be given a series of evidence-based alternative coping strategies for managing trauma-related distress such as anxiety, depression, and PTSD. Participants will be asked to set goals related to utilization of these alternative coping strategies. Participants will then be informed that a trained peer who is part of the research team will follow up with them via text message at the monthly time points to review adherence to their goals and offer support.
  Interventions: Behavioral: Trauma-Informed and Peer-Supported Brief Intervention

INTERVENTIONS:
Behavioral: Standard Brief Intervention — Immediately following completion of the baseline assessment, participants will be texted a link to a secure website which contains the participant's personalized feedback. Personalized feedback is automatically presented via a programming algorithm that is based on the participants baseline survey responses. The personalized feedback component will include a personalized substance use profile, information on peer norms, prior substance-related consequences experienced by the participant, practical costs (e.g., money spent on substances, fees for a DUI), and standard protective behavioral strategies to limit substance-related risk.
  Arms: Standard Brief Intervention
Behavioral: Trauma-Informed and Peer-Supported Brief Intervention — In addition to the components of the standard brief intervention, the TIPS-BI will include personalized feedback about participants use of substances to cope. Additionally, participants will be provided with psychoeducation about the link between substance use, trauma, and coping motives, and information highlighting the iatrogenic effects that substance use has on negative emotions. Participants will also be given a series of evidence-based alternative coping strategies for managing trauma-related distress such as anxiety, depression, and PTSD. Participants will be asked to set goals related to utilization of these alternative coping strategies. Participants will then be informed that a trained peer who is part of the research team will follow up with them via text message at the monthly time points to review adherence to their goals and offer support.

SUMMARY:
This proposal seeks to improve a mobile-based brief intervention for young adults who engage in heavy alcohol use and have experienced interpersonal trauma. The enhancement involves incorporating adaptive coping strategies to address trauma-related distress and engaging peer coaches following the intervention to support sustained treatment effects. Participants will be randomly assigned to receive either the enhanced intervention with peer coaching or a standard version of the brief intervention. Follow-up assessments will be conducted at 3 and 6 months after the intervention. The research team expects that the trauma-informed and peer-supported brief intervention (TIPS-BI) will have low dropout rates, be well-received by participants, and lead to greater reductions in alcohol use than the standard brief intervention.

DETAILED DESCRIPTION:
Alcohol is the most commonly used substance in the United States, with emerging adults (EAs) showing the highest rates of heavy use among all age groups. Persistent heavy drinking in this population is linked to a range of negative outcomes, including poor mental health, reduced life satisfaction, cognitive impairments, academic difficulties, increased risk for motor vehicle accidents, and the development of substance use disorders.

Brief interventions (BIs) for substance use typically involve one or two individual sessions that provide personalized feedback. These interventions aim to challenge inaccurate normative beliefs and emphasize personal consequences of substance use. While BIs have demonstrated success in reducing alcohol consumption and related problems in numerous clinical trials, their impact is often limited. Common challenges include small effect sizes that diminish over time and reduced effectiveness among individuals with interpersonal trauma-specifically, trauma involving human-perpetrated violence and associated emotional distress.

One explanation for these limited outcomes is that BIs are not tailored to high-risk groups such as trauma survivors. Improving BIs may require addressing two key gaps: (1) targeting coping motives-strong predictors of heavy and persistent drinking among trauma-exposed individuals that are typically not addressed in standard BIs, and (2) incorporating peer coaches to support continued gains after the intervention.

There are compelling reasons to integrate trauma content, coping strategies, and peer support into BIs for substance-using EAs. Emerging adulthood is the developmental stage with the highest risk of experiencing interpersonal trauma, which is linked to poor mental health, low social support, and elevated alcohol use. Research indicates that coping with negative emotions is a common motive for substance use in this age group-especially among trauma-exposed individuals-yet these connections are not typically addressed in standard BIs. Additionally, traditional BIs often fail to provide adaptive strategies for managing trauma-related emotional distress, despite the availability of evidence-based coping techniques.

Peer influence also plays a critical role in both initiating and maintaining substance use during emerging adulthood. Including affiliated peers in in-person BIs has improved treatment outcomes in past studies. However, few interventions have extended peer involvement to the post-intervention period, despite the demonstrated success of peer coaches in other health domains.

Further, in-person, counselor-delivered BIs have been criticized as costly and difficult to implement broadly, limiting their scalability. Since few EAs actively seek substance use prevention or treatment services, there is a pressing need for low-cost, accessible delivery methods. Given the widespread use of mobile phones, mobile-delivered BIs represent a promising approach. Early evidence suggests they can be effective with EAs, though engagement tends to be low. Incorporating peer coaches into follow-up may help address this issue and boost engagement.

The primary aim of the proposed study is to evaluate the feasibility and efficacy of a mobile-delivered, trauma-informed, and peer-supported brief intervention (TIPS-BI) for emerging adults with a history of interpersonal trauma. This study will advance the BI literature by:

1. including content that links trauma to substance use and teaches emotion regulation strategies, and
2. integrating trained peer coaches into the text-message follow-up phase.

A total of 190 emerging adults (ages 18-29, with 60% expected to be female) who have a history of interpersonal trauma and report recent heavy alcohol use will be enrolled in a two-arm randomized controlled trial. Participants will be assigned to one of two conditions:

Group 1: Mobile-delivered TIPS-BI with peer coach follow-up (N=95)

Group 2: Mobile-delivered standard substance use BI (N=95)

Aim 1: Assess the feasibility and acceptability of the TIPS-BI. The investigators hypothesize that the TIPS-BI will result in low dropout rates (<10%) at follow-up, comparable to the standard BI. They also expect participants to rate the TIPS-BI as satisfactory, relevant, helpful, and minimally burdensome.

Aims 2 & 3: Evaluate the efficacy of the TIPS-BI. It is hypothesized that participants in the TIPS-BI group will show greater reductions in alcohol use and coping motives at 3- and 6-month follow-ups compared to those receiving the standard BI. Additionally, the TIPS-BI is expected to lead to greater improvements in coping self-efficacy at both follow-up time points.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 29
2. Ability to speak and understand English
3. Access to a cell phone
4. Lifetime history of interpersonal trauma exposure
5. Heavy alcohol use

Exclusion Criteria:

1) Currently receiving psychological therapy or psychotropic medication for substance use.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol use | Change from Baseline to 3-month follow-up
  The Daily Drinking Questionnaire
Alcohol use | Change from Baseline to 6-month follow-up
  The Daily Drinking Questionnaire
Alcohol consequences | Change from Baseline to 3-month follow-up
  The Brief Young Adult Alcohol Consequences Questionnaire
Alcohol consequences | Change from Baseline to 6-month follow-up
  The Brief Young Adult Alcohol Consequences Questionnaire
Intervention feasibility | 6-month follow-up
  Percentage of drop out in the interventions
Intervention acceptability | Baseline
  Participants in both the standard and modified brief interventions will be asked to rate on a Likert scale how satisfied they were with the brief intervention content.
Peer coaching acceptability | Baseline
  Participants in the modified brief intervention will be asked to rate on a Likert scale how satisfied they were with the peer coaching.

SECONDARY OUTCOMES:
Alcohol use motives | Baseline to 3-month follow-up
  Modified Drinking Motives Questionnaire - Revised
Alcohol use motives | Baseline to 6-month follow-up
  Modified Drinking Motives Questionnaire - Revised
Substance-related coping | Baseline to 3-month follow-up
  The Brief Cope Inventory; scores range from 2 to 8; higher scores reflected greater use of the specified coping method
Substance-related coping | Baseline to 6-month follow-up
  The Brief Cope Inventory; scores range from 2 to 8; higher scores reflected greater use of the specified coping method
Coping self-efficacy | Change from baseline to 3-month follow-up
  The Coping Self-Efficacy Scale; scores range from 0-260; higher scores reflect greater coping self-efficacy.
Coping self-efficacy | Change from baseline to 6-month follow-up
  The Coping Self-Efficacy Scale; scores range from 0-260; higher scores reflect greater coping self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Western Kentucky University, Bowling Green, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonomo Y, Coffey C, Wolfe R, Lynskey M, Bowes G, Patton G. Adverse outcomes of alcohol use in adolescents. Addiction. 2001 Oct;96(10):1485-96. doi: 10.1046/j.1360-0443.2001.9610148512.x. PMID 11571067
- [Background] Wilk AI, Jensen NM, Havighurst TC. Meta-analysis of randomized control trials addressing brief interventions in heavy alcohol drinkers. J Gen Intern Med. 1997 May;12(5):274-83. doi: 10.1046/j.1525-1497.1997.012005274.x. PMID 9159696
- [Background] Kurtz SP, Pagano ME, Buttram ME, Ungar M. Brief interventions for young adults who use drugs: The moderating effects of resilience and trauma. J Subst Abuse Treat. 2019 Jun;101:18-24. doi: 10.1016/j.jsat.2019.03.009. Epub 2019 Mar 24. PMID 31174710
- [Background] Bountress KE, Cusack SE, Sheerin CM, Hawn S, Dick DM, Kendler KS, Amstadter AB. Alcohol consumption, interpersonal trauma, and drinking to cope with trauma-related distress: An auto-regressive, cross-lagged model. Psychol Addict Behav. 2019 May;33(3):221-231. doi: 10.1037/adb0000457. Epub 2019 Mar 14. PMID 30869917
- [Background] Tanner-Smith EE, Parr NJ, Schweer-Collins M, Saitz R. Effects of brief substance use interventions delivered in general medical settings: a systematic review and meta-analysis. Addiction. 2022 Apr;117(4):877-889. doi: 10.1111/add.15674. Epub 2021 Oct 14. PMID 34647649
- [Background] Teeters JB, Soltis KE, Murphy JG. A Mobile Phone-Based Brief Intervention With Personalized Feedback and Text Messaging Is Associated With Reductions in Driving After Drinking Among College Drinkers. J Stud Alcohol Drugs. 2018 Sep;79(5):710-719. doi: 10.15288/jsad.2018.79.710. PMID 30422784